CLINICAL TRIAL: NCT07387913
Title: Evaluation of the Effect of Leucocyte Platelet-Rich Fibrin (L-PRF) Technique Applied in Post-extraction Sockets Before Placement of Dental Implants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Maria Pavli, BDS(Hons), MSc, PhD candidate, Oral and Maxillofacial University Clinic, Athens Dental School, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 415/23.05.2019
Record Dates: First submitted 2026-01-18; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: L-PRF; Dental Implants; Osseointegration; Alveolar Bone Grafting
Keywords: Dental implant; Platelet-rich fibrin; Alveolar ridge preservation; Dental implant stability; Tooth-socket preservation
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Control (No Intervention): In these post-extraction sockets no intervention takes place.
- Group 2: Allograft and collagen membrane (Experimental): In order to perform alveolar ridge preservation in this group allograft and collagen membrane are placed in the post-extraction sockets.
  Interventions: Procedure: Allograft and collagen membrane
- Group 3: Allograft and L-PRF membrane (Experimental): In order to perform alveolar ridge preservation in this group allograft and L-PRF membrane are placed in the post-extraction sockets.
  Interventions: Procedure: Allograft and L-PRF membrane
- Group 4: L-PRF membrane (Experimental): In order to perform alveolar ridge preservation in this group L-PRF membrane is placed in post-extraction sockets.
  Interventions: Procedure: L-PRF

INTERVENTIONS:
Procedure: Allograft and collagen membrane — The post-extraction sockets will be filled with allograft particles and collagen membrane.
  Other Names: Group 2
  Arms: Group 2: Allograft and collagen membrane
Procedure: Allograft and L-PRF membrane — The post-extraction sockets will be filled with allograft particles and L-PRF membrane.
  Other Names: Group 3
  Arms: Group 3: Allograft and L-PRF membrane
Procedure: L-PRF — The post-extraction sockets will be filled with L-PRF membrane.
  Other Names: Group 4
  Arms: Group 4: L-PRF membrane

SUMMARY:
Aim of study: The application of L-PRF membrane in post-extraction sockets outmatches the use of a) allograft covered with a collagen fleece b) allograft combined with L-PRF membrane c) natural healing, with reference to bone remodeling and regeneration of post-extraction sockets.

Moreover, it will be examined whether the application of L-PRF membrane leads to faster bone maturation and creation of a favorable biological environment for earlier implant placement.

Materials and methods: This study is taking place in Athens University Dental School, in Oral and Maxillofacial Surgery Clinic. All patients participating in the present study received thorough informed consent. All forty patients participating in this study, were subjected in at least one atraumatic and flapless extraction of a single rooted tooth in the maxilla or mandible. Then, the patients were randomly divided in four categories with regards to management of the socket: a) no intervention i.e. Natural healing b) application of L-PRF membrane in the socket c) application of allograft (Phoenix) covered with a collagen fleece d) application of allograft (Phoenix) covered with a L-PRF membrane. Interrupted sutures will be performed for the four extraction socket groups.

Radiographic examination (localized CBCT) was obtained immediately before the extraction, as well as three months post-operatively (localized CBCT) in order to assess the changes in the alveolar ridge dimensions. The next stage of the study refers to the rehabilitation of the edentulous region.

Before each patient was subjected to dental implant placement, a bone biopsy was obtained.

Therefore, all the biopsy specimens obtained went through histological evaluation in order to assess qualitative and quantitative features.

ELIGIBILITY:
Inclusion Criteria:

1. Single-rooted teeth needed to be extracted in the maxilla or mandible
2. Patient in good general health as documented by self-assessment
3. Patients must be committed to the study and sign the informed consent
4. Adults only as participants

Exclusion Criteria:

1. No systemic medical condition that could interfere with the surgical procedure or planned treatment.
2. Smokers >20 cig/day
3. Current pregnancy or breast feeding
4. Radiotherapy or chemotherapy in head and neck area intravenous and oral bisphosphonates or anti-angiogenic drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Radiographic assessment of the bone specimens | 3 months
  Comparison of quantitative clinical alveolar ridge dimensions (in mm) between the four groups will be performed, 3 months after alveolar ridge preservation. Radiographic evaluation will take place and changes in horizontal dimension will be measured. The horizontal bone width of the ridge at the time of the extraction and after 3 months during the implant placement procedure will be measured in mm.

SECONDARY OUTCOMES:
Radiographic assessment of the bone specimens | 3 months
  Comparison of quantitative clinical alveolar ridge dimensions (in mm) between the four groups will be performed, 3 months after alveolar ridge preservation. Radiographic evaluation will take place and changes in vertical dimension will be measured. The vertical bone height of the ridge at the time of the extraction and after 3 months during the implant placement procedure will be measured in mm.
Histological assessment of the bone harvested from the post-extraction sockets | 3 months
  Measure quantitative histologic characteristics of new bone formation between the four groups after 3 months of alveolar ridge preservation by quantifying the distribution in (%) of new vital bone formed at the healed socket site.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Lygidakis, Associate Professor, Study Chair — National and Kapodistrian University of Athens
Locations (1):
- Athens Univeristy Dental School, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choukroun, J., Adda, F., Schoeffler, C., &Vervelle, A. (2001). Une opportunit?? enparo-implantologie: Le PRF. Implantodontie, 42, 55-62.
- [Background] Castro AB, Meschi N, Temmerman A, Pinto N, Lambrechts P, Teughels W, Quirynen M. Regenerative potential of leucocyte- and platelet-rich fibrin. Part B: sinus floor elevation, alveolar ridge preservation and implant therapy. A systematic review. J Clin Periodontol. 2017 Feb;44(2):225-234. doi: 10.1111/jcpe.12658. Epub 2017 Jan 10. PMID 27891638
- [Background] Castro AB, Van Dessel J, Temmerman A, Jacobs R, Quirynen M. Effect of different platelet-rich fibrin matrices for ridge preservation in multiple tooth extractions: A split-mouth randomized controlled clinical trial. J Clin Periodontol. 2021 Jul;48(7):984-995. doi: 10.1111/jcpe.13463. Epub 2021 Apr 18. PMID 33847018
- [Background] Miron RJ, Zucchelli G, Pikos MA, Salama M, Lee S, Guillemette V, Fujioka-Kobayashi M, Bishara M, Zhang Y, Wang HL, Chandad F, Nacopoulos C, Simonpieri A, Aalam AA, Felice P, Sammartino G, Ghanaati S, Hernandez MA, Choukroun J. Use of platelet-rich fibrin in regenerative dentistry: a systematic review. Clin Oral Investig. 2017 Jul;21(6):1913-1927. doi: 10.1007/s00784-017-2133-z. Epub 2017 May 27. PMID 28551729
- [Background] Temmerman A, Vandessel J, Castro A, Jacobs R, Teughels W, Pinto N, Quirynen M. The use of leucocyte and platelet-rich fibrin in socket management and ridge preservation: a split-mouth, randomized, controlled clinical trial. J Clin Periodontol. 2016 Nov;43(11):990-999. doi: 10.1111/jcpe.12612. Epub 2016 Sep 21. PMID 27509214
- [Background] Vignoletti F, Matesanz P, Rodrigo D, Figuero E, Martin C, Sanz M. Surgical protocols for ridge preservation after tooth extraction. A systematic review. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:22-38. doi: 10.1111/j.1600-0501.2011.02331.x. PMID 22211304
- [Background] Barone A, Ricci M, Tonelli P, Santini S, Covani U. Tissue changes of extraction sockets in humans: a comparison of spontaneous healing vs. ridge preservation with secondary soft tissue healing. Clin Oral Implants Res. 2013 Nov;24(11):1231-7. doi: 10.1111/j.1600-0501.2012.02535.x. Epub 2012 Jul 12. PMID 22784417
- [Background] Dohan Ehrenfest DM, Pinto NR, Pereda A, Jimenez P, Corso MD, Kang BS, Nally M, Lanata N, Wang HL, Quirynen M. The impact of the centrifuge characteristics and centrifugation protocols on the cells, growth factors, and fibrin architecture of a leukocyte- and platelet-rich fibrin (L-PRF) clot and membrane. Platelets. 2018 Mar;29(2):171-184. doi: 10.1080/09537104.2017.1293812. Epub 2017 Apr 24. PMID 28437133
- [Background] Cammack GV 2nd, Nevins M, Clem DS 3rd, Hatch JP, Mellonig JT. Histologic evaluation of mineralized and demineralized freeze-dried bone allograft for ridge and sinus augmentations. Int J Periodontics Restorative Dent. 2005 Jun;25(3):231-7. PMID 16001735